CLINICAL TRIAL: NCT00547131
Title: A Pilot Feasibility Study of Intracerebral Microdialysis to Determine the Neuropharmacokinetics of Temozolomide
Brief Title: Temozolomide in Treating Patients With Primary Brain Tumors or Metastatic Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 05117; P30CA033572 (NIH); CHNMC-05117; CDR0000570280 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Brain and Central Nervous System Tumors; Metastatic Cancer
Keywords: tumors metastatic to brain; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — Temozolomide; Chromatography, Liquid; Mass Spectrometry; Radiosurgery

INTERVENTIONS:
Drug: temozolomide
Other: laboratory biomarker analysis
Other: liquid chromatography
Other: mass spectrometry
Other: pharmacological study
Procedure: conventional surgery
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Collecting fluid samples through a catheter may help doctors find out how well temozolomide spreads throughout the brain.

PURPOSE: This clinical trial is studying temozolomide in treating patients with primary brain tumors or metastatic brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of microdialysis for assessing the intracerebral distribution of temozolomide in patients with primary or metastatic brain tumors.
* Determine the interstitial pharmacokinetics of temozolomide using an intracerebral microdialysis catheter in these patients.
* Determine the feasibility of assessing brain tumor metabolism using a microdialysis catheter to measure intracerebral levels of glucose, lactate, pyruvate, glutamate, and glycerol in these patients.

OUTLINE: Patients are assessed for viable tumor during a debulking craniotomy or stereotactic biopsy. If viable tumor is confirmed, patients undergo placement of an intracerebral microdialysis (MD) catheter. The catheter, which is perfused continuously over 24 hours with artificial cerebrospinal fluid, is placed directly into the residual brain tumor or peritumoral brain tissue for neuropharmacokinetic studies of temozolomide. At least 25 hours but no more than 72 hours after placement of the catheter, patients receive a single dose of oral temozolomide. At the same time, intracerebral MD is initiated and serial samples of dialysate (i.e., brain extracellular fluid [ECF]) are collected periodically over 24 hours for analysis of intracerebral concentrations of temozolomide by liquid chromatography/tandem mass spectrometry. Serial blood samples for measuring plasma levels of temozolomide are also drawn and plasma temozolomide levels are compared with those in the brain ECF. Additional ECF samples are obtained to assess biochemical markers of brain tumor metabolism (i.e., glucose, lactate, pyruvate, glutamate, or glycerol) at least one hour before and 24 hours after administration of temozolomide.

After completion of study therapy, patients are followed for up to 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a primary or metastatic brain tumor for which temozolomide would be an appropriate chemotherapy treatment postoperatively
* Disease requires a debulking craniotomy or a stereotactic biopsy to diagnose or differentiate between tumor progression and treatment-induced effects after radiotherapy with or without chemotherapy

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 2.0 mg/dL
* AST ≤ 4 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 time ULN
* Mini Mental Status Exam score ≥ 15
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No allergy to temozolomide
* No serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No concurrent chemotherapy or radiotherapy during the period of time that the microdialysis catheter is placed intracerebrally and until it is removed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence rate of clinically symptomatic intratumoral hemorrhage
Incidence rate of CNS infection
Incidence rate of catheter malfunction

SECONDARY OUTCOMES:
Systemic and intracerebral pharmacokinetic profile of temozolomide using a microdialysis catheter

CONTACTS AND LOCATIONS:
Overall Officials: Jana Portnow, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California